CLINICAL TRIAL: NCT02245802
Title: Multicenter Prospective Validation Study on the Prediction of In-hospital Mortality Using CU Prediction Model for Patients With Bleeding Peptic Ulcers
Brief Title: Multicenter Validation on Predicting Mortality for Patients With Bleeding Peptic Ulcers
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Tokyo University (Other); National Taiwan University Hospital (Other); Tsuyama Central Hospital, Okayama (Unknown); Hiroshima City Asa Hospital, Hiroshima (Unknown); Mitoyo General Hospital (Unknown); Okayama University (Other)
Responsible Party: Principal Investigator, Philip Wai Yan Chiu, Professor, Department of Surgery, Institute of Digestive Disease, Chinese University of Hong Kong
Other Study IDs: CRE-2010.207
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Bleeding Peptic Ulcer
Keywords: Bleeding peptic ulcer; Prediction model; Mortality; Prediction of in-hospital mortality for bleeding peptic ulcer
MeSH Terms: conditions — Peptic Ulcer Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low risk group: CU Prediction model < 3
- High risk group: CU Prediction model >=3

SUMMARY:
This study aimed to validate CU prediction model on mortality for patients with high risk bleeding peptic ulcers after therapeutic endoscopy.

DETAILED DESCRIPTION:
Despite advances in management of patients with bleeding peptic ulcers, mortality is still 10%. We previously reported a prediction score for ulcer bleeding related mortality developed from a local cohort. The risk factors for mortality included patients older than 70, presence of co-morbidity, more than one listed co-morbidity, hematemesis, SBP < 100 mmHg, in-hospital bleeding, rebleeding, and need for surgery.

Study objective This study aimed to validate the prediction of mortality among patients with bleeding peptic ulcers from different Asian countries.

Method Consecutive patients with bleeding peptic ulcers who presented to the study centers in Hong Kong, Japan and Taiwan were recruited after successful primary endoscopic hemostasis. The baseline demographics, ulcer characteristics, the predictive factors, 30 days mortality, rebleeding, hospital stay and need of surgery were recorded. The accuracy of prediction for adverse events including mortality and rebleeding with the prediction risk scoring system would be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presented with bleeding peptic ulcers
2. Age > 18 year old
3. Informed consent for the study and OGD

Exclusion Criteria:

1. Unable or refuse to give consent
2. Onset more than 7 days
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bleeding peptic ulcers who required endoscopic therapy
Sampling Method: Non-Probability Sample
Enrollment: 785 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Accuracy in prediction of peptic ulcer bleeding related mortality | 30 days
  The CU prediction score would be calculated from addition of all the risk factors scores. . The calculated predictive score collected from the whole group of patients would be analyzed using the receiver operating characteristic (ROC) curve and represented using the area under curve (AUC). An AUC of 0.5 would be interpreted as poor predictive power whereas a value of 1.0 would indicate excellent predictive power.

SECONDARY OUTCOMES:
Mortality difference between high risk and low risk group | 30 days
Need of Surgery | 30 days
Need of Transfusion | 30 days
  Need of transfusion as represented by number of units transfused
Complication rate | 30 days
Hospital stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chiu, MD, Principal Investigator — Department of Surgery, The Chinese University of Hong Kong
Locations (1):
- Combined Endoscopy Center, Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Background] Chiu PW, Ng EK, Cheung FK, Chan FK, Leung WK, Wu JC, Wong VW, Yung MY, Tsoi K, Lau JY, Sung JJ, Chung SS. Predicting mortality in patients with bleeding peptic ulcers after therapeutic endoscopy. Clin Gastroenterol Hepatol. 2009 Mar;7(3):311-6; quiz 253. doi: 10.1016/j.cgh.2008.08.044. Epub 2008 Sep 13. PMID 18955161